CLINICAL TRIAL: NCT03747354
Title: Serum (PLR), (LMR), (MPV) and (NLR) in Behcet Disease and Their Correlation With Disease Activity
Brief Title: Assessment of Disease Activity in Behcet by Complete Blood Count
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, esraa omar ali, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: disease activity in behcet
Record Dates: First submitted 2018-11-11; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complete blood count (Active Comparator): blood samples will be taken from patient and complete blood count is done early morning
  Interventions: Diagnostic Test: blood samples
- erythrocyte sedimentation rate (Active Comparator): blood samples will be taken from patient and erythrocyte sedimentation rate is done
  Interventions: Diagnostic Test: blood samples

INTERVENTIONS:
Diagnostic Test: blood samples — blood samples

SUMMARY:
* To determine platelet to lymphocyte ratio (PLR), lymphocytes to monocytes ratio (LMR), mean platelet volume (MPV) and neutrophile lymphocyte ratio (NLR), levels in Behçet's disease (BD)
* To investigate their correlation with disease activity.

DETAILED DESCRIPTION:
Behçet' s disease (BD) is a complex, inflammatory multisystem disorder characterized by recurrent attacks of oral ulcers, genital ulcers, cutaneous lesions, and inflammatory ocular finding. The vascular inflammatory change is known to be the main histopathology. There is no sensitive or specific laboratory test or pathologic findings , the diagnosis relies heavily on mucocutaneous manifestations and other clinical findings.

In the previous studies,In order to diagnose and monitor disease activity in BD, many cytokines and biomarkers have been identified such as increased blood levels of neopterin, a1-antitrypsin, a2- macroglobulin were correlated with disease activity. Some markers including interleukin-6, -interleukin1b, tumor necrosis factor a (TNF-a), thrombomodulin, E-selectin, vascular endothelial growth factor, antilysozyme(5), serum endocan, serum growth differentiation factor (GDF-15), serum alpha 1-acid glycoprotein, and homocysteine had been considered as inflammatory indicators in BD, However, they are not routinely used in clinical practice as they are not simple or easily derived. Limitations of these markers also include the reflection of short-term inflammatory activity and low discrimination ability with other superimposed inflammatory conditions.

Currently, the platelet to lymphocyte ratio (PLR), lymphocyte to monocyte ratio (LMR), and similar parameters (red blood cell distribution width (RDW), mean platelet volume (MPV) and neutrophil to lymphocyte ratio (NLR), which can be calculated from the peripheral blood easily, have been demonstrated as a new expression of the systemic inflammatory indicators that can aid in the diagnosis and assessment of disease severity in many diseases, such as ankylosing spondylitis,rheumatoid arthritis,systemic lupus erythematosus,and psoriatic Arthritis.nevertheless, only a few studies have investigated RDW, NLR, PLR, or MPV values in patients with BD, none of which have evaluated the role of LMR in BD, not even the relationships between LMR, PLR levels, and disease activity in patients with BD. The mean size of the thrombocytes have been reported on the blood count as mean platelet volume (MPV). MPV is indirectly associated with the activity of platelets. Large platelets are more active than small ones by means of metabolic and enzymatic function. In addition, they also have a higher potential of thrombogenicity. LMR is an easy-to-calculate indicator that can be calculated by leukocyte subgroup of complete blood count. Also, it has been reported that LMR ratio might have prognostic importance for some diseases. Therefore, to better understand these serum inflammatory parameters in BD and to gain deeper insight into the roles of LMR, MPV, NLR and PLR in BD, a prospective study to assess them all together in BD Will conducted

ELIGIBILITY:
Inclusion Criteria:

* -Patient diagnosed as behcet disease by a rheumatologist
* Age from 18 to 70 years old

Exclusion Criteria:

* - Skin diseases,
* Autoimmune diseases,
* Inflammatory or infectious diseases,
* Allergy,
* Subjects with chronic diseases such as cardiovascular disorders, diabetes mellitus, or hematological, kidney, or liver diseases, hypertension, or malignant diseases
* unwilling to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
serum (PLR), (LMR), (MPV) and (NLR) in behcet disease and their correlation with disease activity. | baseline
  * To determine platelet to lymphocyte ratio (PLR), lymphocytes to monocytes ratio (LMR), mean platelet volume (MPV) and neutrophile lymphocyte ratio (NLR), levels in Behçet's disease (BD)
  * To investigate their correlation with disease activity

CONTACTS AND LOCATIONS:
Overall Officials: esraa omar, master, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang Y, Zang M, Li S. Serum PLR and LMR in Behcet's disease: Can they show the disease activity? Medicine (Baltimore). 2017 May;96(21):e6981. doi: 10.1097/MD.0000000000006981. PMID 28538403